CLINICAL TRIAL: NCT05422365
Title: Open, Multicenter, International Study to Evaluate the Efficacy, Safety and Tolerability of Bioven, Manufactured by Biopharma Plasma LLC, in Adult Patients With Chronic Primary Immune Thrombocytopenia (ITP)
Brief Title: Intravenous Immunoglobulin (IVIG, Bioven) Efficacy and Safety in Chronic Primary Immune Thrombocytopenia (ITP) in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Biopharma Plasma LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-BV-ITP-BP
Record Dates: First submitted 2022-06-14; First posted 2022-06-16 (Actual); Results first posted 2024-09-23 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-04

CONDITIONS: Primary Immune Thrombocytopenia
Keywords: IVIG; ITP; immunomodulatory therapy; intravenous immunoglobulin; chronic primary immune thrombocytopenia
MeSH Terms: conditions — Purpura, Thrombocytopenic, Idiopathic | interventions — Immunoglobulins, Intravenous; Solutions

STUDY DESIGN:
Intervention Model Description: Open, multicenter, international, uncontrolled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main Group (Experimental): Patients included in the study will receive the intravenous immunoglobulin (IVIG, Bioven), 10% solution for infusion according to the protocol for the use of IVIG in ITP treatment - at a dose of 0.8-1.0 g / kg once a day for 2 consecutive days, the course dose is 1.6-2.0 g / kg.
  The next day after the administration of the drug, the patient undergoes blood sampling to determine the level of platelets, the level of immunoglobulin G (IgG), and the Coombs test.
  This procedure will also be carried out on days 7, 14, 21, and 28 after the first injection of the drug to monitor the patient's performance.
  Interventions: Drug: Intravenous immunoglobulin (IVIG), 10% solution for infusion

INTERVENTIONS:
Drug: Intravenous immunoglobulin (IVIG), 10% solution for infusion — The study drug is administrated at a dose 0.8-1.0 g / kg once a day for 2 consecutive days, the course dose is 1.6-2.0 g / kg.
  Other Names: Bioven, 10% solution for infusion

SUMMARY:
The study will involve patients with chronic immune thrombocytopenia. This disease is diagnosed in the presence of isolated thrombocytopenia (decrease in platelet count only), except for other reasons. The addition of "chronic" means that the disease lasts more than 12 months.

Patients included in the study will receive Bioven, 10% solution for infusion according to the protocol for the use of IVIG in ITP - at a dose of 0.8-1.0 g / kg 1 time per day for 2 consecutive days, the course dose of 1.6-2.0 g / kg according to the "Guideline on the clinical investigation of human normal immunoglobulin for intravenous administration (IVIG)", rev. 3, 28 June 2018. After administration of the investigational drug, patients will be under medical supervision for 28 days.

The stay of patients in the study - at least 4 weeks.

DETAILED DESCRIPTION:
The investigational drug, IVIG, is used for immunomodulatory therapy in the treatment of autoimmune diseases.

The study will involve patients with chronic immune thrombocytopenia. This autoimmune disease is diagnosed in the presence of isolated thrombocytopenia (decrease in platelet count only), except for other reasons. The addition of "chronic" means that the disease lasts more than 12 months.

Screening stage The patient or her legal representative must sign an informed consent. After the informed consent signing procedure, the patient is screened and assessed for compliance with the inclusion and non-inclusion (exclusion) criteria.

Clinical stage After the patient is included in the study, according to the protocol, he/she is hospitalized and the study drug is administered at a dose of 0.8-1.0 g/kg once a day for 2 days (the course dose is 1.6-2.0 g/kg). The next day after the administration of the drug, the patient undergoes blood sampling to determine the level of platelets, the level of immunoglobulin G (IgG) and the Coombs test. This procedure will also be carried out on days 7, 14, 21 and 28 after the first injection of the drug to monitor the patient's performance.

The final stage The blood sampling procedure to determine the above indicators will be carried out on days 7, 14, 21, and 28 after the first administration of the drug to monitor the patient's performance.

ELIGIBILITY:
Inclusion criteria:

* Signed Patient Informed Consent Form for participation in the study;
* Men and women aged 18-65;
* Confirmed primary chronic ITP (lasting > 12 months since diagnosis);
* A full blood count should be normal except for the isolated thrombocytopenia. Patients with low hemoglobin levels (but above 90 g / l) may be included if there are symptoms of bleeding;
* If bleeding symptoms are diagnosed, the reticulocyte count should be measured;
* Platelet count <30 x 109 / L;
* If the patient is taking corticosteroids, the treatment regimen/dose should be stable (at least 2 weeks prior to screening);
* Negative pregnancy test (for women of child-bearing potential);
* Willingness to use effective and reliable methods of contraception throughout the entire study period;
* The results of physical, instrumental, and laboratory examination of patients should be within the normal range or deviations should be regarded by the researcher as clinically insignificant;
* Ability, according to the researcher, to follow all the requirements of the study protocol;

Exclusion criteria:

* Known intolerance to plasma and immunoglobulin preparations;
* Drug allergy or hypersensitivity to immunoglobulin preparations;
* Confirmed deficiency of immunoglobulin A (IgA) and antibodies to IgA.
* Contraindications to immunoglobulin administration according to the instructions for medical use;
* Pregnancy and lactation;
* Any clinically significant hepatic impairment (increase of serum transaminase levels by more than 3 times the upper limit of normal);
* Serum creatinine levels are more than two times higher than the upper limit of normal for a given age and sex;
* Severe cardiovascular insufficiency (HF III);
* History of thrombosis or presence of significant risk factors for thrombosis.
* Patients with preventive splenectomy;
* Hemostatic disorders other than chronic thrombocytopenia;
* Persons with acute or exacerbation of chronic diseases of the gastrointestinal tract associated with the risk of bleeding, acute infectious diseases, pathologies of the respiratory system;
* Proven case of primary immunodeficiency;
* Secondary immune thrombocytopenia;
* Virus infections (Epstein-Barr, Cytomegalovirus, Parvovirus, Hepatitis B and C);
* Documented HIV infection
* Positive reaction of Wassermann (RW) test result;
* Systemic immunopathological diseases (rheumatic diseases, nephritis, etc.);
* Oncological diseases;
* Diabetes mellitus;
* Thyroid diseases;
* History of mental illness;
* Known drug addiction;
* Any other concomitant decompensated diseases or acute conditions, the presence of which, according to the researcher, may significantly affect the results of the study;
* The need to prescribe drugs that are incompatible with the administration of the drug in this study: other immunoglobulin preparations in addition to the study drug, cytostatic drugs, monoclonal antibodies, Avatrombopag);
* Experimental treatment (e.g. Rituximab therapy) for 3 months prior to screening);
* Blood transfusions or transfusions of blood products in the last 6 months prior to inclusion in the study;
* Administration of IVIG 30 days prior to screening;
* Participation in any other study currently or within the last 30 days;

Criteria for exclusion of subjects (discontinuation of treatment with the study drug):

* Patient's wish
* Occurrence of severe and/or unexpected Adverse events (AE) or Adverse reactions (AR) in patient during the study, that require discontinuation of the drug;
* The need to prescribe drugs prohibited in this study.
* Significant deterioration of the patient's condition during the study period;
* Failure of the patient to adhere to the treatment regimen;
* Failure of the patient to follow the procedures established under the protocol;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- Ukraine (12):
  - Municipal non-profit enterprise "City Clinical Hospital No. 4" of the Dnipro City Council, Dnipro
  - Municipal non-profit enterprise "Khmelnytskyi Regional Hospital" of the Khmelnytskyi Regional Council, Khmelnytskyi
  - Municipal Non-Profit Enterprise "Kirovohrad Regional Hospital of the Kirovohrad Regional Council", Kropyvnytskyi
  - Medical Center "OK!Clinic+" of the Company with Limited Liability "International Institute of Clinical Research", Kyiv
  - Municipal Non-Profit Enterprise of Kyiv Regional Council "Kyiv Regional Oncology Dispensary", Kyiv
  - Municipal non-profit enterprise "Kyiv City Clinical Hospital No. 9" of the executive body of the Kyiv City Council (Kyiv City State Administration), Kyiv
  - "Arensia Exploratory Medicine" Limited Liability Company Medical Center, Kyiv
  - State Institution "Institute of Blood Pathology and Transfusion Medicine of the National Academy of Medical Sciences of Ukraine", Lviv
  - Minicipal enterprise "Rivne regional clinical hospital" of Rivne regional council, Rivne
  - Municipal Non-Profit Enterprise of Sumy Regional Council "Sumy Regional Clinical Hospital", Sumy
  - Municipal non-profit enterprise "Ternopil University Hospital" of Ternopil Regional Council, Ternopil
  - Municipal Non-Profit Enterprise "Zakarpattia Regional Clinical Hospital named after Andriy Novak" of Zakarpattia Regional Council, Uzhhorod

IPD SHARING:
Plan to Share IPD: Yes
The results will be published after trial completion. Access to parts of the Clinical Study Report (CSR) planned after the release of scientific publications.
  Individual participant data (IPD) with the code of each patient will be available In CSR
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After the scientific publication of trial results, 3 months later
Access Criteria: For specialists in field medicine, pharmacy, scientists

REFERENCES:
- See also: Guideline on the clinical investigation of human normal immunoglobulin for intravenous administration (IVIg), rev. 4, 16 December 2021 — https://www.ema.europa.eu/en/documents/scientific-guideline/guideline-clinical-investigation-human-normal-immunoglobulin-intravenous-administration-ivig-rev-4_en.pdf

RESULTS

PARTICIPANT FLOW:
Groups:
- Main Group: Patients included in the study will receive the intravenous immunoglobulin (IVIG, Bioven), 10% solution for infusion according to the protocol for the use of IVIG in ITP treatment - at a dose of 0.8-1.0 g / kg once a day for 2 consecutive days, the course dose is 1.6-2.0 g / kg.
  The next day after the administration of the drug, the patient undergoes blood sampling to determine the level of platelets, the level of immunoglobulin G (IgG), and the Coombs test.
  This procedure will also be carried out on days 7, 14, 21, and 28 after the first injection of the drug to monitor the patient's performance.
  Intravenous immunoglobulin (IVIG), 10% solution for infusion: The study drug is administrated at a dose 0.8-1.0 g / kg once a day for 2 consecutive days, the course dose is 1.6-2.0 g / kg.
Period: Overall Study
Arm/Group | Main Group
Started | 32
Completed | 32
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Main Group
Number analyzed (Participants) | 32
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 32
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 41 [18 to 71]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 7
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ukraine | 26
  Turkey | 6

OUTCOME MEASURES:

1. Primary Outcome: Part (Percent) of Patients With Response (R)
Description: platelet count >30 x 109 /l and at least 2-fold increase of the baseline count, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding
Time Frame: 28 days after first administration of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
Participants | 24

2. Secondary Outcome: Part (Percent) of Patients With Complete Response (CR)
Description: platelet count >100 x 109 /l, confirmed on at least 2 separate occasions at least 7 days apart, and absence of bleeding. Complete response (CR) was achieved in 13 patients during the study.
  CR = 13/32 = 40.63 % (23,61%; 57,64%) This corresponds 40,63% from total number of patients. The confidence interval for this value is 23.61% to 57.64%
Time Frame: 28 days after first administration of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
percentage of participants | 40.63 [23.61 to 57.64]

3. Secondary Outcome: Part (Percent) of Patients With no Response (NR)
Description: platelet count < 30 x 109/L or less than a 2-fold increase of the baseline count. It should be confirmed by at least 2 blood tests or presence of bleeding
Time Frame: 28 days after first administration of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
percentage of participants | 25 [9.99 to 40]

4. Secondary Outcome: Part (Percent) of Patients With Loss of Response (R)
Description: Decreasing platelet count (< 30 x 109/L or less than a 2-fold increase of the baseline count) or development of bleeding. Platelet count should be confirmed at least two times, with an interval of 1 day.
Time Frame: 28 days after first administration of the study drug
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
percentage of participants | 31.25 [15.19 to 47.31]

5. Secondary Outcome: Part (Percent) of Patients With Loss of Complete Response (CR)
Description: decreased platelet count <100 x 109/L or development of bleeding
Time Frame: 28 days after first administration of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Main Group
Number analyzed (Participants) | 13
Participants | 13

6. Secondary Outcome: Time (in Days) From Treatment Start to Response (R)
Description: Time calculated from first infusion (treatment start) to the day when the response (R) criteria are achieved
Time Frame: 28 days after first administration of the study drug
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Main Group
Number analyzed (Participants) | 32
days | 2 [2 to 3]

7. Secondary Outcome: Time (in Days) From Treatment to Complete Response (CR)
Description: Time calculated from first infusion (treatment start) to the day when the complete response (CR) criteria are achieved
Time Frame: 28 days after first administration of the study drug
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Main Group
Number analyzed (Participants) | 32
days | 2 [2 to 4]

8. Secondary Outcome: Duration (in Days) of Response (R)
Description: Time calculated from the day when the complete response (R) criteria are achieved, to the day when loss of complete response (R) criteria is achieved
Time Frame: 28 days after first administration of the study drug
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Main Group
Number analyzed (Participants) | 24
days | 27 [25 to 29]

9. Secondary Outcome: Duration (in Days) of Complete Response (CR)
Description: Time calculated from the day when the complete response (CR) criteria are achieved, to the day when loss of complete response (CR) criteria are achieved
Time Frame: 28 days after first administration of the study drug
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Main Group
Number analyzed (Participants) | 13
days | 19 [13 to 25]

10. Other Pre Specified Outcome: Frequency (Percent) of Adverse Events
Description: Part of the drug administration cases with adverse events, from all cases of study drug administration
Time Frame: 28 days after first administration of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
Participants | 4

11. Other Pre Specified Outcome: Frequency of Serious Adverse Events
Description: Part of the drug administration cases with serious adverse events, from all cases of study drug administration
Time Frame: 28 days after first administration of the study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Main Group
Number analyzed (Participants) | 32
Participants | 1

ADVERSE EVENTS:
Time Frame: 28 days
Description: Definitions of adverse events is similar to clinicaltrials.gov
Arm/Group | Main Group
All-Cause Mortality (participants affected / at risk) | 0/32
Serious Adverse Events (participants affected / at risk) | 1/32
Other Adverse Events (participants affected / at risk) | 4/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Group (N=32)
Vein thrombosis (Blood and lymphatic system disorders) | 1 (1) — Thrombosis of superficial vein of right leg
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Main Group (N=32)
Headache (Nervous system disorders) | 3 (3)
Allergic reaction (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-07-03): https://cdn.clinicaltrials.gov/large-docs/65/NCT05422365/Prot_SAP_000.pdf